CLINICAL TRIAL: NCT03270969
Title: Pharmacokinetics of Tenofovir Disoproxil Fumarate/Emtricitabine for HIV Pre-exposure Prophylaxis in Transgender Women Receiving Feminizing Hormone Therapy
Brief Title: A Pharmacokinetic Evaluation of Tenofovir/Emtricitabine as HIV Pre-Exposure Prophylaxis in Transgender Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0491-17-FB
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Tenofovir; Emtricitabine; emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TDF/FTC (Experimental): Tenofovir Disoproxil Fumarate/Emtricitabine group HIV-uninfected transgender women receiving feminizing hormone therapy plus tenofovir disoproxil fumarate/emtricitabine
  Interventions: Drug: Tenofovir Disoproxil Fumarate/Emtricitabine

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate/Emtricitabine — Participants will receive daily TDF/FTC for 14 days
  Other Names: Descovy and Truvada

SUMMARY:
Human immunodeficiency virus (HIV) persists worldwide as an immense health burden among vulnerable populations. HIV pre-exposure prophylaxis (PrEP) has offered the promise of limiting the global burden of HIV. The objective of this proposal is to conduct a pharmacokinetic (PK) study in transgender women to describe the pharmacokinetics of tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) as PrEP within this population.

DETAILED DESCRIPTION:
PrEP is a critical component of comprehensive transgender medical care. The proposed open-label, intensive PK study will inform the pharmacologic impact of combining PrEP and concurrent feminizing hormone regimens. The investigators hypothesize transgender women will achieve similar PrEP concentrations compared to the historical controls, and that hormone concentrations (estrogen and testosterone) will not be affected. The aims of this study are to (1) to determine if concurrent use of TDF/FTC as PrEP in combination with feminizing hormones alters the PK of tenofovir (TFV) and FTC and (2) to determine if concurrent use of PrEP with feminizing hormones alters serum estradiol and testosterone concentrations. To achieve these aims, this study will enroll transgender women who are receiving either oral/sublingual or transdermal estradiol with spironolactone. Using intensive PK sampling, plasma and intracellular TDF/FTC concentrations will be measured after 14 days of oral TDF/FTC.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Self identify as a transgender woman.
* Receiving estradiol (oral/sublingual tablets or transdermal patches) with oral spironolactone for at least 3 months prior to study entry.
* Serum estradiol level >100 pg/mL.
* Non-reactive 4th or 5th generation screening test for HIV.
* Adults (19 years or older).
* Able to read and speak English to ensure appropriate ability to obtain informed consent.

Exclusion Criteria:

* Participants will not be included in the study if one, or more, of the following criteria are met:
* Use of drugs known to be contraindicated with TDF, FTC, estradiol, or spironolactone within 30 days of study entry. The study team will review all concomitant medications at screening based on the US Department of Health and Human Services drug interaction table and the drug product labeling.
* Use of injectable estradiol (valerate or cypionate).
* Presence of any active condition or clinically significant disease that, in the investigator's opinion, would compromise the subject's safety or outcome of the study, including qualifying for non-occupational post-HIV exposure prophylaxis.
* Signs or symptoms of acute HIV infection within the last 30 days.
* Laboratory values obtained within 30 days prior to study entry:
* Creatinine clearance (CrCl) less than 60 mL/min as estimated by the Cockcroft-Gault equation.
* Positive hepatitis B surface antigen and/or hepatitis C antibody.
* Alanine transaminase (ALT), Aspartate transaminase (AST) or alkaline phosphatase > 5x the upper limit of normal (ULN).
* Hemoglobin <10 g/dL.
* Platelets <50,000/mm3.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender women
Enrollment: 15 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
TFV plasma exposure | 14 days
  Intensive PK sampling compared to historical controls

SECONDARY OUTCOMES:
FTC plasma exposure | 14 days
  Intensive PK sampling compared to historical controls
Tenofovir-diphosphate (TFV-DP) intracellular concentrations | 14 days
  Peripheral blood mononuclear cells (PBMC) concentrations compared to historical control
Emtricitabine-triphosphate (FTC-TP) intracellular concentrations | 14 days
  Peripheral blood mononuclear cells (PBMC) concentrations compared to historical control
TFV maximum plasma concentration (Cmax) | 14 days
  Cmax of TFV compared to historical control
FTC maximum plasma concentration (Cmax) | 14 days
  Cmax of FTC compared to historical control
Estradiol serum concentrations | 14 days
  Before and after intervention
Testosterone serum concentrations | 14 days
  Before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Scarsi, PharmD, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Cirrincione LR, Podany AT, Havens JP, Bares SH, Dyavar SR, Gwon Y, Johnson TM, Amoura NJ, Fletcher CV, Scarsi KK. Plasma and intracellular pharmacokinetics of tenofovir disoproxil fumarate and emtricitabine in transgender women receiving feminizing hormone therapy. J Antimicrob Chemother. 2020 May 1;75(5):1242-1249. doi: 10.1093/jac/dkaa016. PMID 32065631